CLINICAL TRIAL: NCT00176046
Title: Prospective Controlled Randomized Feasibility Study on a Treatment With Viscum Album in Patients With Breast Cancer to Identify Appropriate Surrogate Parameters for a Randomized Study of the Efficacy of Treatment With Mistletoe Extracts
Brief Title: Mistletoe Extract in Early or Advanced Breast Cancer, A Feasibility Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Heidelberg University (Other)
Collaborators: Verein für Krebsforschung, Arlesheim, Swizzerland (Unknown); Weleda AG, D-73525 Schwäbisch Gmünd (Unknown)
Responsible Party: Principal Investigator, Cornelia von Hagens, Head Complementary & Integrative Medicine, Dep. 4.2, Heidelberg University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WD 40
Record Dates: First submitted 2005-09-10; First posted 2005-09-15 (Estimated); Last update posted 2017-05-08 (Actual); Status verified 2009-06

CONDITIONS: Metastatic Breast Cancer
Keywords: breast cancer; mistletoe; complementary therapy; quality of life; immune function; breast cancer (UICC stage I/II)
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- viscum album pini (Experimental): immediate start of treatment with Iscador P s.c.
  Interventions: Drug: viscum album pini
- waiting group (Active Comparator): identical treatment with Iscador P s.c. after waiting period of 3 months
  Interventions: Drug: viscum album pini

INTERVENTIONS:
Drug: viscum album pini — s.c. injection of 0,001-20 mg 3 times per week
  Other Names: Iscador P serie 0, 1, 2
  Arms: viscum album pini
Drug: viscum album pini — s.c. injection 0,001-20 mg 3 times per week
  Other Names: Iscador P Serie 0, 1, 2
  Arms: waiting group

SUMMARY:
The purpose of this feasibility study is to identify appropriate surrogate parameters for a randomized study to examine the efficacy of a complementary therapy with an extract of viscum album (Iscador P) in patients with breast cancer.

DETAILED DESCRIPTION:
The study consists of three parts. Part 1 is a prospective non-randomized feasibility study in patients with breast cancer after primary surgery during chemotherapy or endocrine therapy comparing blood count, lymphocytes, quality of life and local and general side effects between the groups Part 2 is a prospective randomized feasibility study with a waiting list for three months comparing changes in quality of life, depression, diurnal cortisol profile and expression of zeta-chains in T- and NK-cells after three months of treatment or waiting in patients of two different strata (early breast cancer UICC I/II and metastatic breast cancer) Part 3 consists of two follow-up periods of 12 months respective. Patients may choose to continue, quit or restart mistletoe treatment upon their own decision, endpoints from part 2 are evaluated every 6 months.

ELIGIBILITY:
Inclusion Criteria:

* breast cancer
* desire for additional therapy with mistletoe extracts

Exclusion Criteria:

* contraindication for a therapy with mistletoe extracts(allergy, tuberculosis, hyperthyreosis, acute infectious disease, intracranial pressure in case of tumors or metastasis)
* current medication with glucocorticoids or other immunosuppressive therapies
* other concomitant complementary therapies
* prior therapy with mistletoe extracts > 2 years or during the last 6 months
* karnofsky-Index <60

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 1999-05 (Actual); Primary Completion 2009-06 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
blood count | 6-30 months
lymphocytes | 6-30 months
lymphocyte stimulation | 4 months
quality of life | 6-30 months
anxiety and depression | 6-30 months
diurnal profile of cortisol | 6-30 months
expression of zeta-chains on T- and NK-cells | 6-30 months

SECONDARY OUTCOMES:
local reactions | 6-30 months
documentation of concomitant medication | 6-30 months
documentation of concomitant therapies | 6-30 months

CONTACTS AND LOCATIONS:
Overall Officials: Cornelia U. von Hagens, MD, Principal Investigator — Department of Complementary and Integrative Medicine Women's Hospital, University of Heidelberg
Locations (1):
- Department of Complementary and Integrative Medicine, Heidelberg, Baden-Wurttemberg, Germany